CLINICAL TRIAL: NCT02170350
Title: Use of a Brief Mindful Meditation Practice in Adult Cancer Patients Receiving Radiation Therapy
Brief Title: Brief Mindful Meditation Practice in Improving Quality of Life in Patients With Cancer Undergoing Radiation Therapy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Withdrawn by PI
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 14D.272; 2013-107 (Other: CCRRC); JT 5854 (Other: JeffTrial Number)
Record Dates: First submitted 2014-06-19; First posted 2014-06-23 (Estimated); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Malignant Neoplasm
MeSH Terms: conditions — Neoplasms | interventions — Meditation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Brief mindful meditation practice (Experimental): Patients use brief mindful meditation practice (sitting meditation in which the mind is guided to focus in the present, thinking of your existence, and allowing sensations to arise with an openness and curiosity) over 12 minutes daily for 14 days during radiation therapy.
  Interventions: Procedure: Meditation therapy; Other: Quality-of-life assessment; Other: Questionnaire administration

INTERVENTIONS:
Procedure: Meditation therapy — Use brief mindful meditation practice
  Other Names: Meditation
Other: Quality-of-life assessment — Ancillary studies
  Other Names: Quality of life assessment
Other: Questionnaire administration — Ancillary studies

SUMMARY:
This pilot clinical trial studies how well brief mindful mediation practice works in improving quality of life in patients with cancer undergoing radiation therapy. Brief mindful mediation practice may improve the well-being and quality of life of patients with cancer who are undergoing radiation therapy by increasing levels of mindfulness and reducing stress, anxiety/depression, and fatigue.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To investigate the feasibility of a clinical trial using a brief mindful meditation practice during radiation therapy.

SECONDARY OBJECTIVES:

I. To explore the measurable changes in quality of life, fatigue, and mindfulness while using a brief mindful meditation practice during radiation therapy.

OUTLINE:

Patients use brief mindful meditation practice (sitting meditation in which the mind is guided to focus in the present, thinking of your existence, and allowing sensations to arise with an openness and curiosity) over 12 minutes daily for 14 days during radiation therapy.

After completion of study, patients are followed up 4-12 weeks after completion of radiation therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically proven diagnosis of cancer any stage, based upon the following minimum diagnostic workup: History & physical examination, including documentation of Karnofsky Performance Status of 70 - 100% for at least 60 days prior to study entry
2. Patients who are receiving a course of radiation therapy for curative or adjuvant intent
3. Patient who have reported fatigue moderate or higher fatigue (based on the 0-10 Fatigue scale, a fatigue score of 5 or; see Appendix III) while on radiation treatment
4. The patient must be an adult male or female 18 or older
5. Patient must be capable to read and speak English and provide study specific informed consent prior to study entry
6. No prior history of radiation therapy
7. No history of or current active drug/alcohol dependence
8. No patients being decisionally impaired
9. Patients who have home access to a computer, or compact disc audio player

Exclusion Criteria:

1. Patient is under the age of 18
2. Diagnosis of a non-malignant disease and receiving radiation for a pathological diagnosis that is non-cancer
3. Patient who have reported less than moderate fatigue (based on the 0-10 Fatigue scale, a fatigue score less than 5; see Appendix III)
4. Karnofsky performance status of less than 70% within the last 60 days prior to study
5. Prior history of radiation therapy
6. History of or active drug/alcohol dependence or abuse
7. Decisionally impaired patients
8. No access to a computer, or compact disc audio player
9. Patient who are unable to read and speak English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2014-06-06 (Actual); Primary Completion 2015-07-09 (Actual); Study Completion 2016-08-18 (Actual)

PRIMARY OUTCOMES:
Feasibility measured by the proportion of patients who are adherent, defined as successful completion of the course of home base brief mindful meditation practice (at least 8 out of 14 days) and completion of questionnaires at all time points | Up to 12 weeks after completion of radiation therapy
  The portion of patients who complete the brief mindful meditation practice intervention and questionnaires will be computed, along with a one-sided 95% exact confidence interval.

SECONDARY OUTCOMES:
Changes in quality of life assessed by Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) | Baseline to up to 12 weeks after completion of radiation therapy
  Will be analyzed using mixed-effects linear regression. Average changes and associated 95% confidence intervals will be estimated from these models.
Changes in fatigue assessed by FACIT-F | Baseline to up to 12 weeks after completion of radiation therapy
  Will be analyzed using mixed-effects linear regression. Average changes and associated 95% confidence intervals will be estimated from these models.
Changes in mindfulness assessed by Freiburg Mindfulness Inventory | Baseline to up to 12 weeks after completion of radiation therapy
  Will be analyzed using mixed-effects linear regression. Average changes and associated 95% confidence intervals will be estimated from these models.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Werner-Wasik, MD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: Thomas Jefferson University Hospitals — http://www.JeffersonHospital.org